CLINICAL TRIAL: NCT04146948
Title: Comparing Activity of Accessory Inspiratory Muscles and Upper Limb Muscles During Performing Activities of Daily Living Between Patients With Chronic Obstructive Pulmonary Disease and Healthy Adults
Brief Title: The Differences of Muscle Activity Between Patients With COPD and Healthy Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-108-273
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: activities of daily living; accessory inspiratory muscles; oxygen consumption; minute ventilation volume
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- COPD group: No intervention 40 years or older, clinical diagnosis of COPD (Global Initiative for Chronic Obstructive Lung Disease stages I to IV)
  Interventions: Other: no intervention
- healthy group: 40 years or older, not with the clinical diagnosis of COPD
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention in this study

SUMMARY:
The purpose of this study attempts to investigate the differences and relationships of respiratory parameters, muscle activity, and dyspnea during ADL between patients with COPD and age-matched healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* With the clinical diagnosis of COPD

Exclusion Criteria:

* With the clinical diagnosis of asthma or cancer
* With cardiovascular, musculoskeletal and neurological diseases limiting physical activities in daily life
* In the unstable medical state
* MMSE under 25
* Barthel index score under 61

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with COPD will be recruited from the Department of Internal Medicine in National Cheng Kung University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing device | baseline
  The machine analyze the breath of participants including oxygen consumption and minute ventilation volume. Oxygen consumption is reported in mL/min and minute ventilation volume is reported in L/min.
Surface electromyography device | baseline
  The surface EMG is performed to assess the maximum voluntary contraction and muscle activity of upper limb muscles and accessory inspiratory muscles during performing simulated ADL tasks. The maximal voluntary contraction (MVC) is used as the reference level of muscle activity to normalize the EMG data of performing simulated ADL tasks. The muscle activity is reported in percentage.
The clinical Chronic Obstructive Pulmonary Disease questionnaire | baseline
  This is a self-reported questionnaire to measure the impact of COPD on participants' health status. The rating scores is a 7-point scale (0=no limitation, 6=totally limited).Higher scores mean the more severe impact of COPD on participants' daily living.
Modified Borg Scale | baseline
  This is a self-reported scale to measure how much participants perceive dyspnea. The range from 0 which means no difficulty to breathe to 10 which means with maximal difficulty to breathe.
Modified Medical Research Council | baseline
  This is a five-point scale to assess the severity of breathlessness.

SECONDARY OUTCOMES:
EQ-5D questionnaire | baseline
  This is a self-reported questionnaire for measuring generic health status

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

REFERENCES:
- [Derived] Chen CY, Hsu CH, Tsai SH, Lin CF, Lin YC, Hsu HY, Chen CZ, Kuo LC. Association Between Muscle Activity of Upper Limbs and Respiratory Parameters During Functional Performance in People With Chronic Obstructive Pulmonary Disease. Occup Ther Int. 2025 Mar 25;2025:3023322. doi: 10.1155/oti/3023322. eCollection 2025. PMID 40171139